CLINICAL TRIAL: NCT02156557
Title: Phase 1B Study of KCC Peptide Application in the Colon
Brief Title: Study of KCC Peptide Application in the Colon
Acronym: KCC 1B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Danielle Kim Turgeon (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Sponsor-Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HUM00086259
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Colon Polyps; Colorectal Cancer; Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peptide application (Experimental): Investigational Agent Administration
  * KCCFPAQ-GGGSK-(5-FITC)-NH2
  * 1.2 mg lyophilized powder per single-use amber vial
  * Lyophilized powder reconstituted with 10 mL of 0.9% NaCl
  * Final concentration of 76.4 μM for single, one-time topical application
  * The entire 10 mL solution will be sprayed topically onto area of interest by the Clinical Research Associate (CRA)/physician during the procedure through a standard endoscopy spray catheter (Olympus Medical, Tokyo Japan, PW-5V-1)
  Interventions: Biological: Colon KCC Heptapeptide

INTERVENTIONS:
Biological: Colon KCC Heptapeptide — * Your colonoscopy will happen as it would normally, including the medications, the colonoscope, and any clinically indicated biopsies or polypectomies.
  * The fluorescent peptide will be sprayed on to the walls of your colon around the areas that might have a polyp, areas of IBD, or another area of interest. Your doctor will select one area to apply the peptide in your colon. The peptide comes in a single-use sealed vial from the investigational pharmacy. Sterile saline (salt-water) is added to the vial. The powder is mixed well and pulled into a syringe. The peptide is then "injected" into a special, single-use "sprayer", like a garden hose, that fits down the endoscope channel. The peptide will be sprayed in your colon. This is part of the study.
  * The endoscopist will take pictures of the area before and after the peptide spraying. They will use the camera that is part of the colonoscope.
  * We will obtain copies of your endoscopy report and any pathology reports.

SUMMARY:
We are studying new ways to look for abnormal areas/tissues of the colon during a colonoscopy. The current scopes used for colonoscopies are very good. But if the area doesn't look different to the naked eye, then the scope can't improve on that. We are using special stains or dyes and special scopes to see abnormal areas that are hard to see with the naked eye. The stain or dye is "fluorescent", meaning it glows when special light is used in the colonoscopy scope.

You are being asked to let us spray a peptide with a fluorescent tag onto your colon. Peptides are small chains of amino acids (the building blocks that make up proteins) linked together. The peptide we use has 7 amino acids attached to a fluorescent tag ("FIT C" or Fluoresceinisothiocyanate). FITC is used by eye doctors to examine your eyes (the yellow eye drops).

We are testing this "fluorescent peptide" to see if it will stick if there are any abnormal areas. If the peptide "sticks", it will "glow" when a special light in the scope is used. In this study, we will apply the fluorescent peptide to your colon by using a spray tube that fits in the colonoscope.

This is a phase IB study. This means that although we have applied the peptide to 25 people in our first research study, we still need to learn more about "fluorescent peptide" in people. The Food and Drug Administration (FDA) has not approved this agent, but is allowing us to test it in this study. The main goal of this study is to see if the peptide "glows" well and if we can take pictures of areas that do glow.

This is a research study of the peptide and our ability to see it "glow or fluoresce". Being in this study and applying the peptide won't change how our biopsies are taken or how your colonoscopy is done.

ELIGIBILITY:
Inclusion Criteria:

* Subjects felt to be at increased risk for CRC and colonic polyps

OR

-Subjects with known colonic adenomas scheduled for colonic resection

OR

* Subjects who are scheduled for outpatient colonoscopy for follow up surveillance of IBD with known dysplasia or who are at high risk for high grade dysplasia.
* Subjects who are scheduled for outpatient colonoscopy in the medical procedures unit at the University of Michigan Health Center
* All subjects who are medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities) who meet the inclusion/exclusion criteria will be included. Standard practice guidelines for safely proceeding with the procedure will be sufficient for our study
* Adults aged 18 to 100 years
* Willing and able to sign informed consent
* The effects of Colon KCC Heptapeptide (5-FITC-labeled peptide) on the developing human fetus are unknown. For this reason, women of childbearing potential must have a negative pregnancy test on the day of the procedure prior to receiving the Colon KCC Heptapeptide (5-FITC-labeled peptide agent) or be post-menopausal. Post-menopausal women are defined as post-hysterectomy, or over 40 and at least 18 months without menses and not on birth-control.

Exclusion Criteria:

* Subjects with known allergy or negative reaction to fluorescein or derivatives.
* Subjects on active chemotherapy or radiation treatment
* Pregnant or trying to conceive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Validation of binding of peptide | One time during colonoscopy
  The peptide will be applied during colonoscopy to areas that appear abnormal with white light endoscopy. The peptide fluorescence will be assessed via imaging to assess specificity of binding as compared to standard of care pathology interpretation of tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Joshi BP, Dai Z, Gao Z, Lee JH, Ghimire N, Chen J, Prabhu A, Wamsteker EJ, Kwon RS, Elta GH, Stoffel EM, Pant A, Kaltenbach T, Soetikno RM, Appelman HD, Kuick R, Turgeon DK, Wang TD. Detection of Sessile Serrated Adenomas in the Proximal Colon Using Wide-Field Fluorescence Endoscopy. Gastroenterology. 2017 Apr;152(5):1002-1013.e9. doi: 10.1053/j.gastro.2016.12.009. Epub 2016 Dec 22. PMID 28012848